CLINICAL TRIAL: NCT05212948
Title: A Phase 3, Randomized, Observer-Blind, Placebo- Controlled Cross-over Study to Evaluate the Efficacy, Safety, and Immunogenicity of S-268019 for the Prevention of COVID-19
Brief Title: A Study of S-268019 for the Prevention of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2126U0232
Record Dates: First submitted 2022-01-24; First posted 2022-01-28 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — S-268019-b COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-268019-b, Then Placebo (Experimental): Participants will first receive a dose of S-268019-b via intramuscular (IM) injection on Day 1 and Day 29 during the initial vaccination period. After the initial vaccination period, participants will then receive a placebo IM injection (matching S-268019-b) on Day 225 and Day 253.
  Interventions: Drug: S-268019-b; Drug: Placebo
- Placebo, Then S-268019-b (Experimental): Participants will first receive a dose of placebo IM injection (matching S-268019-b) on Day 1 and Day 29 during the initial vaccination period. After the initial vaccination period, participants will then receive S-268019-b IM injection on Day 225 and Day 253.
  Interventions: Drug: S-268019-b; Drug: Placebo

INTERVENTIONS:
Drug: S-268019-b — Solution for IM injection
Drug: Placebo — Saline solution for IM injection

SUMMARY:
The main purpose of this study is to assess the efficacy of S-268019-b for the prevention of COVID-19 in the initial vaccination period prior to crossover in participants without evidence of infection before vaccination as compared to placebo.

DETAILED DESCRIPTION:
Eligible participants will be randomized to receive either S-268019-b or placebo first and then will be crossed over to receive the opposite intervention. The study will consist of two treatment periods, an initial vaccination period (Day 1 to Day 224), and a crossover vaccination period (Day 225 to Day 435).

ELIGIBILITY:
Inclusion Criteria:

* Agree not to participate in any other SARS-CoV-2 prevention trial during the study follow-up.
* Capable of using Diary without difficulties (if applicable, with assistance by caregiver).

Exclusion Criteria:

* Current or history of a laboratory-confirmed diagnosis of SARS-CoV-2 infection or COVID-19.
* Unstable current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disease that, in the opinion of the investigator or subinvestigator, would constitute a safety concern or confound data interpretation.
* Immunosuppression (immunodeficiency, acquired immunodeficiency syndrome [AIDS], use of systemic steroids, use of immunosuppressants within the past 6 months prior to the first dose of study intervention, treatment for malignant tumors, other immunosuppressive therapy).
* Previous vaccination against SARS-CoV-2.
* Any inactivated vaccine received within 14 days prior to the first dose of study intervention.
* Any live vaccine received within 28 days prior to the first dose of study intervention.
* Immunoglobulin preparations, blood products, or a blood transfusion within 3 months prior to the first dose of study intervention.

Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9902 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Buon Ma Thuot City Medical Center, Buon Ma Thuot, Dak Lak, Vietnam

REFERENCES:
- [Result] Dinh Thiem V, Van Anh PT, Van Men C, Hung DT, Pollard AJ, Kamitani A, Tada Y, Fukuyama H, Iwasaki Y, Ariyasu M, Sonoyama T. A SARS-CoV-2 recombinant spike protein vaccine (S-268019-b) for COVID-19 prevention during the Omicron-dominant period: A phase 3, randomised, placebo-controlled clinical trial. Vaccine. 2024 Jun 20;42(17):3699-3709. doi: 10.1016/j.vaccine.2024.04.084. Epub 2024 May 10. PMID 38734495

RESULTS

PARTICIPANT FLOW:
Groups:
- S-268019-b Then Placebo: Participants received a dose of S-268019-b via intramuscular injection on Day 1 and Day 29 during the Initial Vaccination Period. After the Initial Vaccination Period, participants received placebo via intramuscular injection (matching S-268019-b) on Day 225 and Day 253, during the Crossover Vaccination Period.
- Placebo Then S-268019-b: Participants received a dose of placebo via intramuscular injection (matching S-268019-b) on Day 1 and Day 29 during the Initial Vaccination Period. After the Initial Vaccination Period, participants received S-268019-b via intramuscular injection on Day 225 and Day 253, during the Crossover Vaccination Period.
Period: Initial Vaccination Period
Arm/Group | S-268019-b Then Placebo | Placebo Then S-268019-b
Started | 6600 | 3302
Received At Least 1 Dose Of Study Drug (Full Analysis Set (FAS)) | 6581 | 3285
Modified Intent to Treat (mITT) | 5596 | 2805
Immunogenicity Subset | 64 | 34
Completed (Only deaths indicated as leading to study discontinuation are reported in the Participant Flow section. All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section.) | 5315 | 2602
Not Completed | 1285 | 700
Not completed — Withdrawal by Subject | 409 | 199
Not completed — Suspected Pregnancy | 1 | 0
Not completed — Pregnancy | 20 | 14
Not completed — Physician Decision | 686 | 401
Not completed — Lost to Follow-up | 106 | 42
Not completed — Death | 23 | 18
Not completed — Coronavirus Disease 2019 (COVID-19) | 4 | 3
Not completed — Adverse Event | 36 | 23
Period: Crossover Vaccination Period
Arm/Group | S-268019-b Then Placebo | Placebo Then S-268019-b
Started | 5315 | 2602
Received At Least 1 Dose Of Study Drug | 5150 | 2502
Safety Analysis Set (SAS) | 6581 | 3285
Completed (Only deaths indicated as leading to study discontinuation are reported in the Participant Flow section. All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section.) | 5123 | 2503
Not Completed | 192 | 99
Not completed — Withdrawal by Subject | 95 | 57
Not completed — Pregnancy | 6 | 1
Not completed — Physician Decision | 49 | 24
Not completed — Lost to Follow-up | 23 | 8
Not completed — Death | 10 | 5
Not completed — Adverse Event | 9 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of the study intervention during the Initial Vaccination Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | S-268019-b Then Placebo | Placebo Then S-268019-b | Total
Number analyzed (Participants) | 6581 | 3285 | 9866
Age, Customized [Number; unit: Participants]
  <30 years old | 1863 | 954 | 2817
  ≥30 to <40 years old | 1559 | 717 | 2276
  ≥40 to <50 years old | 1194 | 616 | 1810
  ≥50 to <60 years old | 1017 | 521 | 1538
  ≥60 to <65 years old | 418 | 215 | 633
  ≥65 years old | 530 | 262 | 792
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2151 | 1131 | 3282
  Male | 4430 | 2154 | 6584
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 5 | 23
  Not Hispanic or Latino | 6552 | 3269 | 9821
  Unknown or Not Reported | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 6569 | 3275 | 9844
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 9 | 19
anti-Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) N-protein Antibody Test [Count of Participants; unit: Participants] — Positive = evidence of past or present SARS-CoV-2 infection. Negative = no evidence of past or present SARS-CoV-2 infection. Population: Participants in the Full Analysis Set (FAS) missing baseline N-protein antibody data have been excluded.
  Participants
    number analyzed (Participants) | 6535 | 3269 | 9804
    Positive | 816 | 409 | 1225
    Negative | 5719 | 2860 | 8579

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 Reverse Transcription Polymerase Chain Reaction (RT-PCR)-Positive Symptomatic COVID-19 With Onset at Least 14 Days Following Second Vaccination During the Initial Vaccination Period
Description: Participants without evidence of infection before vaccination (that is, seronegative and PCR-negative at baseline) were determined to have symptomatic COVID-19 when at least 1 protocol-specified COVID-19-related symptom and a positive RT-PCR test result were confirmed by the medical monitor within at least 14 days following the second vaccination. RT-PCR testing was based upon nasopharyngeal swab sampling at protocol-specified timepoints.
Time Frame: From Day 43 (14 days after the second dose administration) to Day 224
Population: Modified Intent to Treat (mITT) population: all participants who received at least 1 dose of the study intervention in the Initial Vaccination Period, excluding participants who had evidence of past or present SARS-CoV-2 infection at baseline. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure. Only data collected during the Initial Vaccination Period reported for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- S-268019-b: Participants received a dose of S-268019-b via intramuscular injection on Day 1 and Day 29 during the Initial Vaccination Period.
- Placebo: Participants received a dose of placebo via intramuscular injection (matching S-268019-b) on Day 1 and Day 29 during the Initial Vaccination Period.
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 5156 | 2595
Participants | 323 | 239
Statistical Analysis 1: Comparison: S-268019-b vs Placebo; Vaccine efficacy was calculated with its 95% confidence interval and defined as 1 minus the relative risk (S-268019-b versus placebo), which included the intervention group, baseline age (continuous) as factors as well as the log of the follow-up time as an offset; Test type: Other — Vaccine Efficacy; p = 0.2409, Poisson Regression Model — One-sided P-value was calculated to test the null hypothesis, vaccine efficacy ≤30%; Robust Error Variance; Efficacy = 34.2, 95% CI 2-sided [21.9 to 44.6]

2. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 RT-PCR-Positive Severe COVID-19 in the Initial Vaccination Period With Onset at Least 14 Days Following Second Vaccination
Description: For participants without evidence of infection before vaccination (that is, seronegative and PCR-negative at baseline) who were confirmed to have symptomatic COVID-19 within at least 14 days following the second vaccination, the investigator evaluated if the maximum intensity during the course of the disease met protocol-specified criteria for severe COVID-19.
Time Frame: From Day 43 (14 days after the second dose administration) to Day 224
Population: Modified Intent to Treat (mITT): participants who received at least 1 dose of study drug, excluding participants who had evidence of past or present SARS-CoV-2 infection at baseline. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure. Only data collected during the Initial Vaccination Period reported for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 5181 | 2617
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 RT-PCR-Positive Symptomatic COVID-19 in the Initial Vaccination Period
Description: Participants without evidence of infection before vaccination (that is, seronegative and PCR-negative at baseline) were determined to have symptomatic COVID-19 when at least 1 protocol-specified COVID-19-related symptom and a positive RT-PCR test result were confirmed by the medical monitor. RT-PCR testing was based upon nasopharyngeal swab sampling at protocol-specified timepoints.
Time Frame: Up to Day 224
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 5595 | 2805
Participants | 457 | 313

4. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 RT-PCR-Positive Severe COVID-19 in the Initial Vaccination Period
Description: For participants without evidence of infection before vaccination (that is, seronegative and PCR-negative at baseline) who were confirmed to have symptomatic COVID-19, the investigator evaluated if the maximum intensity during the course of the disease met the protocol-specified criteria for severe COVID-19.
Time Frame: Up to Day 224
Population: Modified Intent to Treat (mITT): participants who received at least 1 dose of study drug, excluding participants who had evidence of past or present SARS-CoV-2 infection at baseline. Only data collected during the Initial Vaccination Period reported for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 5596 | 2805
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 RT-PCR-Positive Symptomatic COVID-19 in the Initial Vaccination Period Regardless of Serostatus or PCR Status at Baseline With Onset at Least 14 Days Following Second Vaccination
Description: A participant was determined to have symptomatic COVID-19 when at least 1 protocol-specified COVID-19-related symptom and a positive RT-PCR test result were confirmed by the medical monitor within at least 14 days following the second vaccination. RT-PCR testing was based upon nasopharyngeal swab sampling at protocol-specified timepoints.
Time Frame: From Day 43 (14 days after the second dose administration) to Day 224
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of the study intervention during the Initial Vaccination Period. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure. Only data collected during the Initial Vaccination Period reported for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 6023 | 3012
Participants | 331 | 242

6. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 RT-PCR-Positive Severe COVID-19 in the Initial Vaccination Period With Onset at Least 14 Days Following Second Vaccination Regardless of Serostatus or PCR Status at Baseline
Description: For participants confirmed to have symptomatic COVID-19 within at least 14 days following the second vaccination, the investigator evaluated if the maximum intensity during the course of the disease met the protocol-specified criteria for severe COVID-19.
Time Frame: From Day 43 (14 days after the second dose administration) to Day 224
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 6049 | 3034
Participants | 0 | 1

7. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 RT-PCR-Positive Symptomatic COVID-19 in the Initial Vaccination Period Regardless of Serostatus or PCR Status at Baseline
Description: A participant was determined to have symptomatic COVID-19 when the participant had at least 1 protocol-specified COVID-19-related symptom and a positive RT-PCR test result confirmed by the medical monitor. RT-PCR testing was based upon nasopharyngeal swab sampling at protocol-specified timepoints.
Time Frame: Up to Day 224
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 6579 | 3285
Participants | 479 | 324

8. Secondary Outcome: Number of Participants With First Occurrence of SARS-CoV-2 RT-PCR-Positive Severe COVID-19 in the Initial Vaccination Period Regardless of Serostatus or PCR Status at Baseline
Description: For participants confirmed to have symptomatic COVID-19, the investigator evaluated if the maximum intensity during the course of the disease met the protocol-specified criteria for severe COVID-19.
Time Frame: Up to Day 224
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of the study intervention during the Initial Vaccination Period. Only data collected during the Initial Vaccination Period reported for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 6581 | 3285
Participants | 0 | 1

9. Secondary Outcome: Number of Participants With First Occurrence of Asymptomatic SARS-CoV-2 Infection in the Initial Vaccination Period
Description: For participants without evidence of infection before vaccination (that is, seronegative and PCR-negative at baseline), asymptomatic SARS-CoV-2 infection was defined as having a positive result of anti-SARS-CoV-2 N-protein antibody test beginning 14 days following the second vaccination and not meeting the protocol-specified criteria of symptomatic COVID-19. Antibodies to SARS-CoV-2 N-protein were used to determine both natural infection and the incidence of asymptomatic infection acquired during the initial vaccination period of the study.
Time Frame: From Day 43 (14 days after the second dose administration) to Day 224
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 5156 | 2595
Participants | 2543 | 1345

10. Secondary Outcome: Percentage of Participants Experiencing Solicited Systemic Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs were defined as the AEs that occurred within the first 7 days after each vaccination and were classified as one of the following: fever, nausea/vomiting, diarrhea, headache, fatigue, and myalgia. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 224
Population: Safety Analysis Set (SAS): all randomized participants who received at least 1 dose of study intervention. Only data collected during the Initial Vaccination Period reported for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 6581 | 3285
Percentage of Participants | 32.7 [31.5 to 33.8] | 23.4 [22.0 to 24.9]

11. Secondary Outcome: Percentage of Participants Experiencing Solicited Local Adverse Events
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited local AEs were defined as the AEs that occurred within the first 7 days after each vaccination and were classified as one of the following: pain, erythema/redness, induration, and swelling. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 224
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 6581 | 3285
Percentage of Participants | 37.7 [36.5 to 38.9] | 14.6 [13.4 to 15.8]

12. Secondary Outcome: Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Antibody
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody level against SARS-CoV-2 was measured by a live virus neutralization assay. The GMT was calculated by taking the back transformation of the arithmetic mean of log-transformed titers. The 95% confidence interval was calculated based on the Student's t distribution of the log-transformed values, then back transformed to the original scale.
Time Frame: Day 57
Population: Immunogenicity Subset: participants who received at least 1 dose of study drug, excluding participants with evidence of past or present SARS-CoV-2 infection at baseline, and had a valid immunogenicity test result prior to the first vaccination dose and at least 1 valid result after the first vaccination dose. 'Overall Number of Participants Analyzed' are participants evaluable for this outcome measure. Only data collected during the Initial Vaccination Period reported for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 58 | 28
Titer | 34.66 [27.04 to 44.41] | 2.69 [2.31 to 3.14]

13. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Neutralizing Antibody
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody level against SARS-CoV-2 was measured by a live virus neutralization assay. The GMFR was calculated by taking the back transformation of the arithmetic mean of the change from baseline in log-transformed titers. The 95% confidence interval was calculated based on the Student's t distribution of the change from baseline in the log-transformed values, then back transformed to the original scale.
Time Frame: Day 57
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 58 | 28
Fold Rise | 13.86 [10.82 to 17.76] | 1.08 [0.92 to 1.25]

14. Secondary Outcome: Seroconversion Rate of SARS-CoV-2 Neutralizing Antibody
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody level against SARS-CoV-2 was measured by a live virus neutralization assay. Seroconversion was defined as a 4-times or higher from baseline in SARS-CoV-2 neutralizing antibody titer, where titer values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Seroconversion rate was defined as the percentage of participants that underwent seroconversion. The 95% confidence interval was calculated using the Clopper-Pearson method.
Time Frame: Day 57
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 58 | 28
Percentage of Participants | 93.1 [83.3 to 98.1] | 3.6 [0.1 to 18.3]

15. Secondary Outcome: GMT of Anti-SARS-CoV-2 S-protein Immunoglobulin G (IgG) Antibody
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The serum neutralizing antibody level against SARS-CoV-2 (anti-spike protein IgG antibody) was measured by a chemiluminescence immunoassay. The GMT was calculated by taking the back transformation of the arithmetic mean of log- transformed titers. The 95% confidence interval was calculated based on the Student's t distribution of the log-transformed values, then back transformed to the original scale.
Time Frame: Day 57
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 58 | 28
Titer | 25209.25 [17163.57 to 37026.44] | 6.39 [3.10 to 13.19]

16. Secondary Outcome: GMFR of Anti-SARS-CoV-2 S-protein IgG Antibody
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The anti-spike protein IgG antibody was measured by a chemiluminescence immunoassay. The GMFR was calculated by taking the back transformation of the arithmetic mean of the change from baseline in log-transformed titers. The 95% confidence interval was calculated based on the Student's t distribution of the change from baseline in the log-transformed values, then back transformed to the original scale.
Time Frame: Day 57
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 57 | 28
Fold Rise | 6710.95 [4556.29 to 9884.54] | 1.46 [0.75 to 2.85]

17. Secondary Outcome: Seroconversion Rate of Anti-SARS-CoV-2 S-protein IgG Antibody
Description: Blood samples for immunogenicity assessments were collected during protocol-specified study visits. The anti-spike protein IgG antibody was measured by a chemiluminescence immunoassay. Seroconversion was defined as a 4-times or higher from baseline in anti-spike protein IgG antibody titer, where titer values reported as below the LLOQ are replaced by 0.5*LLOQ and titer values reported as above the upper limit of quantification (ULOQ) are imputed at the ULOQ value. Seroconversion rate was defined as the percentage of participants that underwent seroconversion. The 95% confidence interval was calculated using the Clopper-Pearson method.
Time Frame: Day 57
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | S-268019-b | Placebo
Number analyzed (Participants) | 57 | 28
Percentage of Participants | 98.2 [90.6 to 100.0] | 7.1 [0.9 to 23.5]

ADVERSE EVENTS:
Time Frame: Day 1 (Baseline) through Day 435
Description: All reported safety data based upon Safety Analysis Set: all randomized participants who received at least 1 dose of study intervention. Safety data presented per pre-specified analysis plan. All deaths regardless of causality or whether they were reported as a reason for study discontinuation or as a serious adverse event are reported in the All-Cause Mortality section. Only deaths indicated as leading to study discontinuation are reported in the Participant Flow section.
Groups:
- S-268019-b: Participants received a dose of S-268019-b via intramuscular injection on Day 1 and Day 29 during the Initial Vaccination Period and then on Day 225 and Day 253 during the Crossover Vaccination Period.
- Placebo: Participants received a dose of placebo via intramuscular injection (matching S-268019-b) on Day 1 and Day 29 during the Initial Vaccination Period and then on Day 225 and Day 253 during the Crossover Vaccination Period.
Arm/Group | S-268019-b | Placebo
All-Cause Mortality (participants affected / at risk) | 29/9083 | 29/8435
Serious Adverse Events (participants affected / at risk) | 154/9083 | 136/8435
Other Adverse Events (participants affected / at risk) | 3647/9083 | 1548/8435
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | S-268019-b (N=9083) | Placebo (N=8435)
Pneumonia (Infections and infestations) | 8 | 9
COVID-19 (Infections and infestations) | 8 | 7
Appendicitis (Infections and infestations) | 4 | 2
Bronchitis (Infections and infestations) | 5 | 4
Tuberculosis (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 1 | 3
Abscess limb (Infections and infestations) | 2 | 0
Rickettsiosis (Infections and infestations) | 2 | 0
Dengue fever (Infections and infestations) | 1 | 1
Encephalitis (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Lung abscess (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fallopian tube abscess (Infections and infestations) | 0/2978 | 1/2781 — Adverse event affected only female participants.
Febrile infection (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Shigella infection (Infections and infestations) | 1 | 0
Dengue haemorrhagic fever (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 1/2978 | 0/2781 — Adverse event affected only female participants.
Bacterial infection (Infections and infestations) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2978 | 1/2781 — Adverse event affected only female participants.
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2978 | 1/2781 — Adverse event affected only female participants.
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Goitre (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Calcium deficiency (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Alcoholic psychosis (Psychiatric disorders) | 3 | 1
Completed suicide (Psychiatric disorders) | 2 | 2
Schizophrenia (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 2
Alcohol use disorder (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Epilepsy (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 1
Cerebrovascular disorder (Nervous system disorders) | 1 | 1
Chorea (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Sciatic nerve neuropathy (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Cataract subcapsular (Eye disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 2 | 4
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 4 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Heart valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 3
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2/2978 | 2/2781 — Adverse event affected only female participants.
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0/2978 | 1/2781 — Adverse event affected only female participants.
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/2978 | 1/2781 — Adverse event affected only female participants.
Ovarian cyst (Reproductive system and breast disorders) | 0/2978 | 1/2781 — Adverse event affected only female participants.
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 1
Death (General disorders) | 9 | 3
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Multi-organ disorder (General disorders) | 2 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 3
Multiple injuries (Injury, poisoning and procedural complications) | 4 | 4
Soft tissue injury (Injury, poisoning and procedural complications) | 3 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 2
Wound (Injury, poisoning and procedural complications) | 2 | 1
Chest injury (Injury, poisoning and procedural complications) | 2 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Venom poisoning (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrical burn (Injury, poisoning and procedural complications) | 1 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Nasal injury (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S-268019-b (N=9083) | Placebo (N=8435)
Headache (Nervous system disorders) | 1235 | 446
Myalgia (Musculoskeletal and connective tissue disorders) | 1029 | 255
Pain (General disorders) | 1689 | 290
Fatigue (General disorders) | 1405 | 468
Injection site pain (General disorders) | 923 | 219
Pyrexia (General disorders) | 676 | 185

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PIs center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 45 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT05212948/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT05212948/SAP_001.pdf